CLINICAL TRIAL: NCT06155435
Title: Effect of Solution-oriented Approach Training for Nulliparous Pregnant Women on Their Traumatic Perception of Chilbirth, Vaginal Birth Self-efficacy and Mode of Birth Choice.
Brief Title: Effect of Solution-focused Approach Training on Traumatic Birth Perception, Vaginal Birth Self-efficacy, Birth Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Tugba Yazıcı Topcu, specialist midwife, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KTU-SABE-TYT-01
Record Dates: First submitted 2023-11-19; First posted 2023-12-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Birth; Self Efficacy; Perception, Self
Keywords: pregnancy; self efficacy; solution-oriented approach training; traumatic birth perception; vaginal birth
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Intervention Model Description: The experimental group was given solution-oriented training
Who Masked: Participant
Masking Description: There was one-way blinding in the randomization of this study. While it is known to the experimental or control class researcher of pregnant women, it can be done by the pregnant woman
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Firstly, the Pregnant Information Form, Traumatic Birth Perception Scale and Vaginal Birth Self-Efficacy Scale forms will be applied.Solution-oriented approach training; It is indicated for pregnant women one by one and in the form of at least 4 entries. A recording will take approximately 30-35 minutes.15-21 days after the solution-oriented approach training is completed the traumatic birth perception and vaginal birth self-efficacy scale form will be applied again.The traumatic birth perception form will be applied again 15-21 days after birth. The woman's birth type will be learned and recorded.
  40 pregnant women will be followed in the experimental group.
  Interventions: Behavioral: solution focused approach training
- control group (No Intervention): Firstly, the Pregnant Information Form, Traumatic Birth Perception Scale and Vaginal Birth Self-Efficacy Scale forms will be applied. will be no intervention on the pregnant women in the control group, and the 15-21st week after the prenatal care given to the pregnant women by the Ministry of Health is completed. Traumatic birth perception and vaginal birth self-efficacy scale form will be filled in on these days. The traumatic birth perception form will be applied again 15-21 days after birth. The woman's birth type will be learned and recorded. 40 pregnant women will be followed in the control group.

INTERVENTIONS:
Behavioral: solution focused approach training — To the woman; A list of education subjects will be sent in order to determine educational changes for birth, birth and postpartum periods. This list will be; It consists of reproductive organs, pregnancy formations, changes, psychological changes, daily life, nutrition, reproductive monitoring, immunization, frequent problems and solution suggestions, danger signs and what to do. Also included in the list are labor, birth cycle, and postpartum periods.
  Other Names: Providing solution-oriented treatment training to pregnant women
  Arms: experimental group

SUMMARY:
Women's psycho-social health during pregnancy could influence the course of pregnancy, psychological and emotional life, not only in labor but also during the postpartum period. Women's perception of birth and their self-efficacy may affect the birth and postpartum period, and their delivery preference. The study aims to examine the effect of solution-oriented approach training on traumatic birth perception, vaginal birth selfefficacy, and delivery preference. It was designed in a randomized controlled experimental type. The sample in the study will comprise 80 pregnant women (40 experimental and 40 control groups) with the help of power analysis. The study is going to be conducted with pregnant women applying to KTU Farabi Hospital between May and December 2022. 6-8 sessions of solution-oriented approach training will be given to pregnant women with 28 weeks of gestation and above and willing to take part in the study, and their delivery preferences will be examined, afterward. The pregnant women in the control group, on the other hand, will not be subjected to any training or interview other than routine pregnancy follow-ups. Data will be gathered through the Pregnant introductory information form, traumatic birth perception scale form, and vaginal birth self-efficacy form. Ethics Committee Permission, institutional permission from the institution where the research will be conducted, and written informed consent from the mothers will be obtained before the research. The data will be statistically evaluated through the SPSS 23 program. Student t-test or Mann-Whitney U tests will be applied for two independent groups. One A Way or Kruskal-Wallis tests will be applied for three or more independent groups, depending on whether the data meet the parametric conditions. Paired T or Wilcoxon tests will be used for two dependent groups, and Friedman or Repeat Measure tests will be applied for three or more groups. In statistical evaluation, p<0.05 will be considered significant.

DETAILED DESCRIPTION:
Pregnancy, birth and postpartum period; It is one of the most special behaviors of women. In this period when the woman plays a very important role after intercourse, her psychological health status can have an impact on her psychological and emotional life, including the course of pregnancy, birth and the period after birth.Sociodemographic characteristics, previous pregnancy or birth history, pregnancy and birth information obtained through hearsay, information obtained from unreliable sources, low health literacy level, not being able to receive adequate and effective prenatal care, and being in your first pregnancy are some of the factors that affect the psychosocial health of women.Although birth, which is the result of pregnancy, is a normal and physiological process, it is one of the unique experiences that affects the woman physically, psychologically and socially and causes significant changes in her life. Although birth is under the influence of all processes of a woman's life, it is especially closely related to how the pregnancy goes and how it is perceived. Although cesarean birth is a preferred method of birth only when vaginal birth is contraindicated or unsafe, this method of birth may be preferred by women for reasons such as the perception of traumatic birth and low self-efficacy for vaginal birth. When we look at the cesarean section rates in live births, it is seen that the total cesarean section rate, which was 48.0% in 2014, increased to 54.4% in 2019 . In our country, where the prenatal care rate is 98%, the fact that cesarean section rates are at such high levels poses a risk for mother-child and public health. Caesarean section birth, which is life-saving in case of medical necessity, increases the maternal morbidity and mortality rate by 2-4 times compared to vaginal births when performed off-label. Also, birth by cesarean section; It poses a risk in situations such as mother-baby bonding, starting and continuing breastfeeding, postpartum recovery and returning to daily life after discharge. Psychosocial and cognitive factors such as a negative past birth experience, negative birth stories, low self-efficacy for vaginal birth, and perceiving birth as traumatic play a role in women's preference for cesarean delivery. In a study conducted with 384 pregnant women in Trabzon province, 56.8% of these pregnant women perceived the birth as moderately traumatic, and 27.1% as highly traumatic. Birth is perceived as traumatic; It may be caused by situations such as fear of birth and low self-efficacy towards birth. Lack of knowledge about birth, labor pain, having a first birth, pain during birth, and inability to cope with the situations encountered cause an increase in the fear of birth and a decrease in birth self-efficacy in these pregnant women. Self-efficacy in birth is defined as "the woman's ability to see in herself the power to cope with the act of birth and her confidence in her abilities". The concept of self-efficacy is a subjective concept, and the level of self-efficacy can also affect the labor process and the fear of birth and therefore the perception of birth as traumatic. Another phenomenon that affects the birth process and the choice of birth method is the "perception of traumatic birth". The perception of traumatic birth is defined as the woman's perception of the birth process as a risk of injury and/or death for herself and her baby. Perception of birth as traumatic can cause depression, increased fear of birth, and negative birth experience in pregnant women.In order for the pregnancy, birth and postpartum period not to deviate from its naturalness and to be completed in a physiologically and psychosocially healthy way, support can be provided to the process through birth preparation classes and various prenatal trainings given to expectant parents. It has been determined that prenatal education given to pregnant women in the third trimester reduces the fear of birth and negative perceptions about birth.The training given to pregnant women by health professionals such as midwives, obstetricians and nurses during the antental period contributes to increasing the pregnant woman's health awareness, increasing her ability to cope with problems related to pregnancy and birth, strengthening her self-efficacy for vaginal birth, and having a positive birth experience. Solution-oriented approach training is of particular importance in helping pregnant women cope with their problems, perceiving pregnancy and birth, and protecting and improving their mental health.Solution-focused approach training is a type of counseling practice called "brief therapy" that was developed under the leadership of Steve de Shazer and Insoo Kim Berg between 1970 and 1980. The aim of this training is to try to solve the individual's basic problems with a short and pragmatic approach and to help the client determine the goal they want to achieve. In solution-focused approach training, unlike classical psychotherapy methods, the focus is on the "solution" instead of the "problem" and the person's past successes, good and strong aspects in his life are emphasized instead of dealing with the problem itself. It focuses on the strengths of the person being trained and the things they want to achieve, and emphasizes that the solution to the problem will come from the person himself and that his self-confidence will increase as a result. In other words, it aims to increase the individual's self-confidence and self-efficacy. One of the most important features of this training is that it provides effectiveness in a short time and lasts 6-10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research
* Being over 20 years old
* Being able to speak Turkish
* Not having any disability such as hearing or vision
* Being nulliparous pregnant
* Being in the 3rd trimester (those who are pregnant between 28-35 weeks)
* Not having received any psychiatric diagnosis before
* No risk of vaginal bleeding, hypertension, diabetes, multiple pregnancy etc. during pregnancy.
* Not having any physical/mental problems that would prevent normal birth.

Exclusion Criteria:

* Pregnant women in high risk groups (arthritis, premature birth, placenta previa, etc.)
* Multigravida pregnant women (pregnant women with 2 or more pregnancies)
* Having received any psychiatric diagnosis and/or receiving psychiatric treatment.

The termination criteria for the cases included in the study will be as follows:

* Intrauterine fetal death during pregnancy,
* Emergence of any risk during pregnancy,

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
traumatic birth perception scale | two months
  It was developed to measure the traumatic birth perception levels of women of reproductive age. There are a total of 13 questions in the scale. These questions; It includes the feelings and thoughts, anxiety, fear and trauma that a woman may experience when she thinks about giving birth. Answers to the questions were scored between 0 and 10, from "none at all" to "most". The total score obtained from the scale shows the level of perception of traumatic birth. The minimum scores that can be obtained from the scale are 0 and the maximum is 130. Total score averages indicate that the 0-26 point range is very low, the 27-52 point range is low, the 53-78 point range is medium, the 79-104 point range is high, and the 105-130 point range indicates that the woman has a very high level of perception of traumatic birth. The Cronbach Alpha reliability coefficient of the scale is 0.895.
vagınal bırth self-effıcacy | two months
  This scale was developed to measure self-efficacy regarding vaginal birth during pregnancy. The scale consists of 9 items and there is an 11-point (0-10) numerical rating scale for each item. Scores range from 0 to 90, with higher scores indicating higher levels of self-efficacy. There are no items in the scale that need to be reverse coded. Cronbach's alpha coefficient, as a reliability criterion to determine the internal consistency of the scale, varies between 0.93 and 0.94.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Teknik Üniversitesi, Trabzon, Turkey (Türkiye)